CLINICAL TRIAL: NCT05767489
Title: Study of Brain Anatomo-functional Substrates Related to the Use of Human Tool by Means of Simultaneous Acquisition of Magnetic Resonance Imaging and Electroencephalogram
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS SYNLAB SDN (Other)
Responsible Party: Sponsor
Other Study IDs: 8/20
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2023-03

CONDITIONS: Patients With Frontal and Parietal Lobe Dysfunction
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: electroencephalogram (EEG) and magnetic resonance (MR) — High-resolution 3D T1 and T2 sequences, acquired in the sagittal plane and MR reconstructed in the remaining orthogonal planes, for morphological assessment of different cortical and subcortical.
  EEG tracing involving recording channels such as eye tracking (eye-tracking: electrooculogram, pupillometry, saccades, fixation times on areas predefined areas), performance measures (response times), electrocardiogram and electromyogram proper to clinical acquisition

SUMMARY:
This is an observational study, conducted on subjects with neurological disorders primarily involving the frontal and parietal lobes of the brain. Throughout the indicated period, the study will aim to enroll 100 subjects divided into 30 units per year. Specifically, the study will be carried out on patients with fronto-parietal dysfunction for whom a prescribed a clinical investigation of electroencephalogram and MRI

ELIGIBILITY:
Inclusion Criteria:

* subjects of either sex with fronto-parietal dysfunction, who are able to able to provide voluntary consent, who have been asked for clinical purposes for an EEG and an MRI

Exclusion Criteria:

* pregnant or presumed pregnant subjects and subjects with claustrophobia or with contraindications to the examination.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with brain dysfunction, particularly affecting the lobe frontal, temporal and parietal
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2025-01-17 (Estimated)

PRIMARY OUTCOMES:
Combination of EEG and functional MR (fMRI) | 1-36 months
  Interception of differences during simultaneous acquisition related to the variation of action readiness (action readiness) suggested by the visual-perceptual context

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Synlab SDN, Naples, Italy

IPD SHARING:
Plan to Share IPD: No